CLINICAL TRIAL: NCT00280241
Title: Phase II Clinical Protocol for the Treatment of Patients With Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: Protocol for the Treatment of Patients With Previously Untreated Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Genentech, Inc. (Industry); Biogen (Industry)
Responsible Party: Principal Investigator, Michael Boyiadzis, Study Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-136
Record Dates: First submitted 2006-01-19; First posted 2006-01-20 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic; Lymphocytic; Leukemia; Fludarabine; Cyclophosphamide; Rituximab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Bronchiolitis Obliterans Syndrome; Leukemia | interventions — fludarabine; Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FLUDARABINE, CYCLOSPHOSPHAMIDE AND RITUXIMAB (Experimental)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Rituximab

INTERVENTIONS:
Drug: Fludarabine — Fludarabine is usually administered by IV infusion over 30 minutes or longer.
Drug: Cyclophosphamide — The dosage is a solution of 20 mg/mI. IV infusion over 1 hour.
Drug: Rituximab — First Infusion: The rituximab solution for infusion should be administered intravenously at an initial rate of 50 mg/hr. Subsequent rituximab infusions can be administered at an initial rate of 100 mg/hr, and increased by 100 mg/hr increments at 30-minute intervals, to a maximum of 400 mg/hr as tolerated.

SUMMARY:
This research study will look at the effects (good or bad) of administering cyclophosphamide, fludarabine, and rituximab. Clinical studies with combination therapy have shown higher response rates than using single drugs, and this study will evaluate the side effects and effectiveness of this combination.

DETAILED DESCRIPTION:
This study is designed to expand on the highly successful combination of rituximab, fludarabine and cyclophosphamide for patients with previously untreated CLL. Responses in the range of 90-98% with 55% complete responses are reported. However, bone marrow toxicity has been a significant problem. This trial is designed to reduce the bone marrow toxicity by decreasing the doses of fludarabine and cyclophosphamide, but doubling the dose of rituximab with a maintenance dose of rituximab for up to two years, to maintain or even enhance efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD20 + CLL
* Peripheral blood absolute lymphocyte count of > 5,000/mm3 obtained within 2 weeks prior to randomization.
* The lymphocytosis must consist of small to moderate size lymphocytes, with ≤55% (no greater than 55%) prolymphocytes, atypical lymphocytes, or lymphoblasts morphologically.
* Phenotypically characterized CD20 + CLL defined as: 1) the predominant population of cells share B-cell antigens with CD5 in the absence of other pan-T-celI markers (CD3, CD2, etc.); 2) B-cell expresses either kappa or lambda light chains; and 3) surface immunoglobulin (slg) with low-cell surface density expression.
* Splenomegaly, hepatomegaly or lymphadenopathy are not required for the diagnosis of CLL.
* Must require chemotherapy. Indications for chemotherapy are one or more of the following:
* One or more of the following disease-related symptoms
* Weight loss >10% within the previous 6 months.
* Fevers of greater than 100.0° F for 2 weeks without evidence of infection.
* Night sweats without evidence of infection.
* Evidence of progressive marrow failure as manifested by the development of or worsening of anemia (< 10 g/dl) and/or thrombocytopenia (< 100,000/mm3).
* Massive (i.e., > 6 cm below left costal margin) or progressive splenomegaly.
* Massive nodes or clusters (i.e., > 10 cm in longest diameter) or progressive
* adenopathy.
* Progressive lymphocytosis with an increase of> 50% over 2 month period, or an anticipated doubling time of less than 6 months.
* NOTE: Marked hypogammaglobulinemia or the development of a monoclonal protein in the absence of any of the above criteria for active disease are not sufficient for protocol therapy.
* Serum creatinine <1.5 mg/dl.
* Bilirubin must be <2 mg/dl, unless secondary to tumor, obtained within 2 weeks prior to randomization.
* Age >18 years.
* Not pregnant (confirmed by serum pregnancy test in females of reproductive potential) or breast feeding, because it is unknown what effect these drugs will have on children.
* ECOG performance status 0-2.
* AST or ATL >2x upper limit of normal unless related to CLL.
* Subject has provided written informed consent.

Exclusion criteria:

* Subjects with autoimmune anemia or thrombocytopenia are not eligible.
* No prior cytotoxic chemotherapy. Patients with a history of steroid treatment for CLL, autoimmune hemolytic anemia, or autoimmune thrombocytopenia are not eligible.
* Subjects with active infections requiring oral or intravenous antibiotics until resolution of the infection and completion of therapeutic antibiotics.
* Women of childbearing potential and sexually active males who refuse to use an accepted and effective method of contraception.
* Subjects with a second malignancy other than basal cell carcinoma of the skin or in situ carcinoma of the cervix are not eligible unless the tumor was treated with curative intent at least two years previously.
* History of HIV
* CNS disease
* History of psychiatric disorder that would make it difficult to enroll and follow the patient on trial.
* New York Heart Classification III or IV heart disease.
* Hepatitis BsAg or Hepatitis C positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2004-06; Primary Completion 2008-02 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Micahel Boyiadzis, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FLUDARABINE, CYCLOSPHOSPHAMIDE AND RITUXIMAB
Started | 65
Completed | 55
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | FLUDARABINE, CYCLOSPHOSPHAMIDE AND RITUXIMAB
Number analyzed (Participants) | 65
Age, Customized [Median (Full Range); unit: years] | 58 [36 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 50

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of Rituximab, Cyclophosphamide and Fludarabine in Patients With Previously Untreated CLL/SLL
Description: The number of patients who experience any grade 3-5 toxicity.
Time Frame: Duration of treatment on study
Measure: Number; unit: participants
Arm/Group | FLUDARABINE, CYCLOSPHOSPHAMIDE AND RITUXIMAB
Number analyzed (Participants) | 65
participants | 42

2. Secondary Outcome: Overall Survival Rate
Description: The percentage of participants who are still alive.
Time Frame: Five years after starting rituximab, cyclophosphamide and fludarabine
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FLUDARABINE, CYCLOSPHOSPHAMIDE AND RITUXIMAB
Number analyzed (Participants) | 65
percentage of participants | 85.5 [73.9 to 92.2]

3. Primary Outcome: Efficacy of Rituximab, Cyclophosphamide and Fludarabine in Patients With Previously Untreated CLL/SLL
Description: The number of patients who experience a complete clinical response.
Time Frame: Three months after the sixth cycle (9 months)
Measure: Number; unit: participants
Arm/Group | FLUDARABINE, CYCLOSPHOSPHAMIDE AND RITUXIMAB
Number analyzed (Participants) | 63
participants | 46

4. Secondary Outcome: Duration of Response
Description: The length of time for which the complete response is maintained.
Time Frame: From complete response to the time of progressive disease, death or last clinical examination
Measure: Median (Full Range); unit: Months
Arm/Group | FLUDARABINE, CYCLOSPHOSPHAMIDE AND RITUXIMAB
Number analyzed (Participants) | 37
Months | 22.3 [5.2 to 42.3]

ADVERSE EVENTS:
Arm/Group | FLUDARABINE, CYCLOSPHOSPHAMIDE AND RITUXIMAB
Serious Adverse Events (participants affected / at risk) | 26/65
Other Adverse Events (participants affected / at risk) | 65/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FLUDARABINE, CYCLOSPHOSPHAMIDE AND RITUXIMAB (N=65)
Hemoglobin (Blood and lymphatic system disorders) | 5
Leukocytes (total WBC) (Investigations) | 7
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 20
Platelets (Investigations) | 2
Blood/Bone Marrow-Other (Blood and lymphatic system disorders) | 1
Supraventricular arrhythmias (SVT/atrial fibrillation/flutter) (Cardiac disorders) | 1
Cardiac-ischemia/infarction (Cardiac disorders) | 2
Edema (General disorders) | 1
Cardiovascular/General-Other (Cardiac disorders) | 1
Prothrombin time (PT) (Blood and lymphatic system disorders) | 1
Rigors, chills (General disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Ileus (or neuroconstipation) (Gastrointestinal disorders) | 1
Infection without neutropenia (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Infection/Febrile Neutropenia-Other (Infections and infestations) | 3
Hypokalemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FLUDARABINE, CYCLOSPHOSPHAMIDE AND RITUXIMAB (N=65)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 7
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 5
Inner ear/hearing (Ear and labyrinth disorders) | 1
Lymphopenia (Investigations) | 1
Hemoglobin (Blood and lymphatic system disorders) | 28
Leukocytes (total WBC) (Investigations) | 41
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 25
Platelets (Investigations) | 25
Blood/Bone Marrow-Other (Blood and lymphatic system disorders) | 1
Edema (General disorders) | 6
Hypotension (Vascular disorders) | 2
Cardiovascular/General-Other (Cardiac disorders) | 2
Hypertension (Vascular disorders) | 2
Fatigue (lethargy, malaise, asthenia) (General disorders) | 53
Weight gain (Investigations) | 2
Weight loss (Investigations) | 3
Constitutional Symptoms-Other (General disorders) | 3
Fever (in the absence of neutropenia, where neutropenia is defined as AGC<1.0 x 10e9/L) (General disorders) | 16
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 12
Rigors, chills (General disorders) | 19
Hot flashes/flushes (Vascular disorders) | 5
Flushing (Vascular disorders) | 2
Injection site reaction (General disorders) | 1
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 10
Erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 1
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 5
Wound-non-infectious (Injury, poisoning and procedural complications) | 2
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 13
Anorexia (Metabolism and nutrition disorders) | 20
Constipation (Gastrointestinal disorders) | 14
Diarrhea (Gastrointestinal disorders) | 15
Dyspepsia/heartburn (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 39
Taste disturbance (dysgeusia) (Gastrointestinal disorders) | 2
Gastrointestinal-Other (Gastrointestinal disorders) | 5
Gastritis (Gastrointestinal disorders) | 1
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 8
Dehydration (Metabolism and nutrition disorders) | 1
Vomiting (Gastrointestinal disorders) | 14
Melena/GI bleeding (Gastrointestinal disorders) | 1
Hemorrhage-Other (Blood and lymphatic system disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
SGOT (AST) (serum glutamic oxaloacetic transaminase) (Investigations) | 3
SGPT (ALT) (serum glutamic pyruvic transaminase) (Investigations) | 3
Alkaline phosphatase (Investigations) | 1
Infection without neutropenia (Infections and infestations) | 23
Infection with unknown ANC (Infections and infestations) | 3
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 2
Wound-infectious (Infections and infestations) | 1
Lymphatics-Other (Blood and lymphatic system disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Muscle weakness (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal-Other (Musculoskeletal and connective tissue disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Memory loss (Nervous system disorders) | 1
Neuropathy - motor (Nervous system disorders) | 6
Neurology-Other (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 15
Dizziness/lightheadedness (Nervous system disorders) | 7
Mood alteration-anxiety, agitation (Psychiatric disorders) | 4
Headache (Nervous system disorders) | 14
Mood alteration-depression (Psychiatric disorders) | 4
Neuropathy-sensory (Nervous system disorders) | 8
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1
Conjunctivitis (Eye disorders) | 1
Vision-blurred vision (Eye disorders) | 3
Ocular/Visual-Other (Eye disorders) | 1
Neuropathic pain (Nervous system disorders) | 1
Pain-Other (General disorders) | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Chest pain (non-cardiac and non-pleuritic) (General disorders) | 2
Abdominal pain or cramping (Gastrointestinal disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 22
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary-Other (Respiratory, thoracic and mediastinal disorders) | 6
Voice changes/stridor/larynx (e.g., hoarseness, loss of voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 1
Dysuria (painful urination) (Renal and urinary disorders) | 2
Urinary frequency/urgency (Renal and urinary disorders) | 4
Creatinine (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes